CLINICAL TRIAL: NCT01816698
Title: A Randomized, Double-Blind, Placebo Control Trial Comparing Effects and Safety of TAURINE GRANULE and Placebo on Blood Pressure in Prehypertensive.
Brief Title: Effects and Safety of Taurine Granule on Blood Pressure in Prehypertensive
Acronym: ESTAB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhiming Zhu (Other)
Responsible Party: Sponsor-Investigator, Zhiming Zhu, Chief Scientist of the National Key Basic Research and Development Program (973 Program), Third Military Medical University
Organization: Third Military Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GZS01167262
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Prehypertension
Keywords: Hypertension; Taurine; Metabolism
MeSH Terms: conditions — Prehypertension; Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Taurine (Active Comparator): Interventions Drug: Taurine granule Arms: Group 1
  Interventions: Drug: Taurine granule
- Placebo (Placebo Comparator): Interventions Drug: Placebo Arms: Group 2
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Taurine granule — 1 package(1.6g taurine granule) once a day after meals, 12 weeks
  Other Names: Taurine granule, H20003861.
  Arms: Taurine
Drug: Placebo — Placebo: 1 package once a day after meals, 12 weeks
  Other Names: Placebo packaged similar to Taurine granule
  Arms: Placebo

SUMMARY:
Prehypertension are associated with an increased risk of atherosclerosis and coronary artery disease, and often complicated with the metabolic disorder of glucose and lipid. The comprehensive prevention of hypertension is still an important and complex clinical issue. Taurine is one of the ingredients of Chinese medicine bezoar ,as an endogenous amino acids is central inhibitory neurotransmitter, can regulate the excitability of nerve tissue, regulate body temperature, therefore, antipyretic, sedative, analgesic, anti-inflammatory,the role of anti-rheumatic, anti-convulsant. In addition, Taurine inhibits platelet aggregation in the circulatory system, lower blood lipids, to maintain the body's normal blood pressure and prevent atherosclerosis; protective effect on myocardial cells, can be anti-arrhythmic; special efficacy to lower blood cholesterol, to treat heart failure. The effect of oral Taurine on blood pressure is not consistent, however, many animal study has shown that oral administration of Taurine, could reduce 24-hour mean arterial systolic and diastolic blood pressure in spontaneous hypertensive rats. Furthermore, Taurine interfere with calcium and low affinity binding of the calcium binding sites, decrease the voltage-dependent Ca2+channel in vascular smooth muscle relaxation, vasodilation, lower blood pressure.In a prospective, double-blind, randomized, and parallel-group study, we will evaluate the effects of Taurine granule on blood pressure and metabolic parameters in prehypertensive and mild hypertensive patients. This study will help develop future comprehensive prevention and treatment strategies for hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Blood pressure: 120mmHg≤SBP<140mmHg.

Exclusion Criteria:

* Diabetes
* Hypertension: SBP≥140mmHg, or DBP≥90mmHg.
* known allergy to trial drugs
* Myocardial infarction or cerebrovascular accident in the year preceding the trial
* Clinical Congestive Heart Failure
* Secondary hypertension
* Pregnancy or lactating women
* Malignant tumor
* Gastroesophageal reflux or gastroduodenal ulcer
* History of hepatitis or cirrhosis
* History of kidney disease
* Body weight﹤35Kg

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The decrease in blood pressure after an 12-week oral Taurine granule administration. | 12 weeks
  Evaluate the effects of Taurine granule on blood pressure and metabolic parameters in prehypertensive patients after an 12-week oral administration.

CONTACTS AND LOCATIONS:
Locations (1):
- The third hospital affiliated to the Third Military Medical University, Chongqing, Chongqing Municipality, China